CLINICAL TRIAL: NCT05930041
Title: The Presence of Injured Submucosal Arteries After Cold Snare Polypectomy(CSP) is Lower Than That of Conventional Hot Snare Endoscopic Mucosal Resection (HS-EMR) for 10-19 mm Nonpedunculated Colorectal Polyps.
Brief Title: Injured Submucosal Arteries After CSP for 10-19 mm Nonpedunculated Colorectal Polyps.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief, Showa Inan General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSP/HSEMR
Record Dates: First submitted 2023-06-25; First posted 2023-07-05 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CSP (Experimental)
  Interventions: Procedure: Experimental CSP
- HS-EMR (Active Comparator)
  Interventions: Procedure: Active Comparator HS-EMR

INTERVENTIONS:
Procedure: Experimental CSP — Either CSP is performed for 10-19 mm nonpedunculated colorectal polyps.
  Arms: CSP
Procedure: Active Comparator HS-EMR — Either HS-EMR is performed for 10-19 mm nonpedunculated colorectal polyps.
  Arms: HS-EMR

SUMMARY:
Cold polypectomy has the advantages of simple operation, less time-consuming and fewer complications. Guidelines have recommended cold snare polypectomy (CSP) to resect small polyps sized <9 mm. CSP was designed to improve the complete resection rate and reduce adverse events. Investigators hypothesize that CSP is better than conventional hot snare endoscopic mucosal resection (HS-EMR) in the presence of injured submucosal arteries detected in the submucosal layer for 10-19 mm nonpedunculated colorectal polyps, resulting in lower delayed bleeding after CSP of 10-19 mm nonpedunculated colorectal polyps.

DETAILED DESCRIPTION:
Cold polypectomy has the advantages of simple operation, less time-consuming and fewer complications. Guidelines have recommended cold snare polypectomy (CSP) to resect small polyps sized <9 mm. CSP was designed to improve the complete resection rate and reduce adverse events. Investigators hypothesize that CSP is better than conventional hot snare endoscopic mucosal resection (HS-EMR) in the presence of injured submucosal arteries detected in the submucosal layer for 10-19 mm nonpedunculated colorectal polyps, resulting in lower delayed bleeding after CS-EMR of 10-19 mm nonpedunculated colorectal polyps. The primary outcome measure was the presence of injured submucosal arteries detected in the submucosal layer. The secondary outcomes included immediate bleeding and the frequency of delayed bleeding requiring endoscopic treatment within 2 weeks after polypectomy. Immediate bleeding was defined as spurting or oozing which continued for more than 30 seconds.

ELIGIBILITY:
Inclusion Criteria:

* at least one polyp sized 10-19 mm (Paris classification Is or IIa) revealed by endoscopic examination.

Exclusion Criteria:

1. American Society of Anesthesiologists status class 3 or above
2. poor bowel preparation (Boston Bowel Preparation Scale <6 points)
3. endoscopic features indicating submucous infiltration or malignancy
4. oral anticoagulants,or antiplatelet agents, or known blood coagulation disorders, or bleeding tendency
5. a history of colorectal resection
6. emergent colonoscopy (haemodynamic instability and/or continued active gastrointestinal bleeding and/or requiring intensive care patients)
7. inflammatory bowel disease, familial polyposis and colorectal cancer
8. pregnancy or lactation
9. severe cardiopulmonary dysfunction, cirrhosis, chronic kidney disease, other malignant tumours or severe infectious diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
the presence of injured submucosal arteries detected in the submucosal layer. | 1 day
  the presence of injured submucosal arteries detected in the submucosal layer.

SECONDARY OUTCOMES:
Delayed bleeding | 14 days
  The frequency of delayed bleeding requiring endoscopic treatment within 2 weeks after polypectomy.
Immediate bleedling | 1 day
  The frequency of Immediate bleeding which was defined as spurting or oozing which continued for more than 30 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General Hospital, Komagane, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kurasawa S, Horiuchi I, Kajiyama M, Kitahara H, Terashima T, Horiuchi A. Injured submucosal arteries following cold snare polypectomy are significantly fewer versus those after endoscopic mucosal resection for 10-19-mm nonpedunculated colorectal polyps. DEN Open. 2025 Mar 18;5(1):e70099. doi: 10.1002/deo2.70099. eCollection 2025 Apr. PMID 40104570